CLINICAL TRIAL: NCT05246709
Title: Randomized Control Study to Evaluate Impact of the Use of Cyanoacrylate Glue on PICC Line Dressing Care in the Infant Cardiac Care Unit at Children's Hospital of New York
Brief Title: Impact of Cyanoacrylate Glue on PICC Line Dressing Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Marianne Garland, Associate Professor of Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAT5997
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Central Line Complication; Neonatal Disease
Keywords: PICC line dressing; cyanoacrylate glue; NICU
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Intervention Model Description: Randomized control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Group (Active Comparator): This group will be received the current standard of care (SOC) dressing method for PICC lines.
  Interventions: Device: Standard transparent film dressing
- Cyanoacrylate Glue Group (Experimental): This group will receive a few drops of cyanoacrylate glue on PICC line site prior to application of usual standard film dressing over the PICC line site.
  Interventions: Device: Cyanoacrylate glue; Device: Standard transparent film dressing

INTERVENTIONS:
Device: Cyanoacrylate glue — Adhesive to be applied on the PICC line site prior to usual standard film dressing over the site, such as SecurePortIV® Catheter Securement Adhesive by Adhezion Biomedical® Cyanoacrylate adhesive that is FDA-approved for securement of vascular access devices.
  Securement method that provides microbial protection by sealing the insertion site.
  Other Names: SecurePortIV® Catheter Securement Adhesive
  Arms: Cyanoacrylate Glue Group
Device: Standard transparent film dressing — A standard transparent polyurethane film dressing, such as 3M TEGADERM Film, for dressing the PICC line area.

SUMMARY:
This study will evaluate whether applying micro drops of cyanoacrylate glue to the participant's peripherally inserted central catheter (PICC) insertion site prior to covering the area of PICC line with a transparent film dressing will make the PICC dressing last longer and prevent an occurrence of PICC line moving out of its original placement. The investigators aims to evaluate whether 1) using the cyanoacrylate glue will lengthen the time to first dressing change; and 2) participants in the experimental arm (glue used) will have fewer dressing changes per week compared to the control arm (standard care) during admission.

DETAILED DESCRIPTION:
The neonatal population poses a unique challenge due to the small surface area of PICC sites, underdeveloped skin layer, and inability to contain the child's movements during a dressing change.

PICC line migration is the most common complication of PICC line maintenance in the neonatal intensive care unit (NICU). Previous studies have found that the PICC migration/dislodgment mostly occurs during PICC dressing changes among the neonatal population.

Recent published studies demonstrated that medical tissue adherence glue, Cyanoacrylate, significantly reduces the incidences of catheter migration and insertion site bleeding of PICC lines in all age of patients including premature infants.

The proposed study is a randomized control study with aimed data collection of 60 participants; of the 60 participants, 50 participants' data are to be used for statistical analysis and additional 10 participants to account for withdrawals.

The participants will be randomly assigned to one of two groups: one (the control group) receiving our standard PICC dressing method and the other (the study group) receiving cyanoacrylate glue at the PICC insertion sites prior to applying a standard transparent film dressing over the PICC sites.

The control group will reflect standard practice of PICC insertion and dressings using a standard transparent polyurethane film dressing, 3M TEGADERM Film.

The study group will reflect the application of a few drops of cyanoacrylate glue, SecurePortIVTM by Adhezion Biomedical® at the insertion sites prior to dressing a PICC line area with a standard transparent polyurethane film dressing.

The aim for this study is to investigate whether the application of cyanoacrylate glue at the insertion sites prior to dressing a PICC line area with a standard dressing will increase the longevity of the PICC line dressing and reduce the incidences of PICC line migration.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the 9 North intensive coronary care unit (ICCU) at NewYork-Presbyterian Morgan Stanley Children's Hospital greater than 35 weeks of corrected gestational age who have a PICC line placed by a NICU provider.

Exclusion Criteria:

* Any patient with a PICC line in situ from an outside hospital.
* Any patient with a PICC line placed by an outside department, namely the interventional radiology department.
* Any patient with a PICC line that is silicon material catheter, such as Vygon Epicutaneo-Cava catheter because of limited accuracy of measuring a movement of the catheter migration after 25 centimeter mark due to absence of a centimeter mark on the catheter.

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2022-02-26 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Garland, MD, Principal Investigator — Morgan Stanley Children's Hospital of NYP
Locations (1):
- NewYork-Presbyterian Morgan Stanley Children's Hospital at CUIMC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to submit the study finding to professional nursing journals, such as Advanced in Neonatal Care, Journal of Neonatal Nursing, and etc
Supporting Information: CSR
Time Frame: 1 to 2 years
Access Criteria: To be determined by the PI

REFERENCES:
- [Background] Acun C, Baker A, Brown LS, Iglesia KA, Sisman J. Peripherally inserted central cathether migration in neonates: Incidence, timing and risk factors. J Neonatal Perinatal Med. 2021;14(3):411-417. doi: 10.3233/NPM-200684. PMID 33459671
- [Background] Bierlaire S, Danhaive O, Carkeek K, Piersigilli F. How to minimize central line-associated bloodstream infections in a neonatal intensive care unit: a quality improvement intervention based on a retrospective analysis and the adoption of an evidence-based bundle. Eur J Pediatr. 2021 Feb;180(2):449-460. doi: 10.1007/s00431-020-03844-9. Epub 2020 Oct 20. PMID 33083900
- [Background] D'Andrea V, Pezza L, Barone G, Pronterà G, Pittiruti M, Vento G. Comparison study: before/after the practice change of the use of medical cyanoacrylate glue for securing ECC (epicutaneo-caval catheter). The Journal of Vascular Access. 2021; 00(0). 1-4.
- [Background] Guido A, Zhang S, Yang C, Pook L. An innovative cyanoacrylate device developed to improve the current standard of care for intravascular catheter securement. J Vasc Access. 2020 May;21(3):293-299. doi: 10.1177/1129729819872881. Epub 2019 Sep 9. PMID 31495268
- [Background] Kleidon TM, Ullman AJ, Gibson V, Chaseling B, Schoutrop J, Mihala G, Rickard CM. A Pilot Randomized Controlled Trial of Novel Dressing and Securement Techniques in 101 Pediatric Patients. J Vasc Interv Radiol. 2017 Nov;28(11):1548-1556.e1. doi: 10.1016/j.jvir.2017.07.012. Epub 2017 Sep 19. PMID 28893464
- [Background] Ostroff M, Zauk A, Chowdhury S, Moureau N, Mobley C. A retrospective analysis of the clinical effectiveness of subcutaneously tunneled femoral vein cannulations at the bedside: A low risk central venous access approach in the neonatal intensive care unit. J Vasc Access. 2021 Nov;22(6):926-934. doi: 10.1177/1129729820969291. Epub 2020 Nov 5. PMID 33148114
- [Background] Sharpe E, Kuhn L, Ratz D, Krein SL, Chopra V. Neonatal Peripherally Inserted Central Catheter Practices and Providers: Results From the Neonatal PICC1 Survey. Adv Neonatal Care. 2017 Jun;17(3):209-221. doi: 10.1097/ANC.0000000000000376. PMID 28045704

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Cyanoacrylate Glue Group
Started | 15 | 17
Completed | 15 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Cyanoacrylate Glue Group | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 8 [6 to 18] | 7 [5 to 11] | 7 [6.0 to 15.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 9 | 8 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Duration of Longevity of PICC Line Dressing
Description: Duration of longevity defined as the number of days the PICC line dressing lasts from the scheduled dressing change.
Time Frame: Up to 7 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control Group | Cyanoacrylate Glue Group
Number analyzed (Participants) | 15 | 17
days | 2 [2 to 3] | 4 [3 to 7]

2. Secondary Outcome: Number of PICC Line Migrations
Description: A PICC line migration is defined as a change in the length of catheter extruding from the insertion site - a catheter migration of more than 0.25 cm will be counted. The reported values represent the total number of PICC line migrations observed across all participants.
Time Frame: Until PICC line removal (approximately 12 weeks)
Measure: Number; unit: PICC line migrations
Arm/Group | Control Group | Cyanoacrylate Glue Group
Number analyzed (Participants) | 15 | 17
PICC line migrations | 6 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Control Group | Cyanoacrylate Glue Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT05246709/Prot_SAP_000.pdf